CLINICAL TRIAL: NCT00706368
Title: Taking Charge of my Health: A Trial to Investigate the Accuracy and Acceptability of Self-Diagnostic Methods for Vaginitis in Adolescent Females
Brief Title: Accuracy and Acceptability of Self-Diagnostic Methods for Vaginitis in Adolescent Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Jill Huppert M.D., MPH, CCHMC Adolescent Medicine Department
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K23AI063182 (NIH); K23AI063182 (NIH)
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-05

CONDITIONS: Trichomonas Vaginalis
Keywords: Sexually transmitted infections; Acceptability; Adolescent vaginitis
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants in this group will perform self-tests for the first half of the study and will have clinical examinations for the second half of the study
  Interventions: Device: Point of care tests
- 2 (Experimental): Participants in this group will have clinical examinations for the first half of the study and will perform self-tests for the second half of the study
  Interventions: Device: Point of care tests

INTERVENTIONS:
Device: Point of care tests — Several point-of-care tests are offered: OSOM TV rapid trichomonas test; OSOM BV Blue rapid test; pHEMalert vaginal pH test. All subjects receive the OSOM TV test, while the other two are optional.

SUMMARY:
Symptoms of vaginitis are common among adolescent females, although studies have shown that neither experienced clinicians nor patients can accurately diagnose the cause of vaginitis based on symptoms alone. The purpose of this study is to investigate the accuracy and acceptability of self-diagnostic methods for vaginitis in adolescent females.

DETAILED DESCRIPTION:
Vaginal symptoms are common among adolescent females. Vaginal symptoms can result from alterations in the normal flora such as candidiasis or bacterial vaginosis (BV), or from sexually transmitted infections (STIs) such as trichomonas vaginalis (Tv). However, studies have shown that neither experienced clinicians or patients can accurately diagnose the etiology of vaginitis based on symptoms alone, and the standard evaluation (pelvic examination and wet mount) has limitations.

As an alternative to the standard evaluation, there are several objective, point-of-care tests that can be performed on vaginal secretions, which could be useful in discriminating between the various causes of vaginitis. These include a rapid test for trichomonas vaginalis, a rapid test for bacterial vaginosis, and the vaginal pH and amine test. The aims of this study are to explore the feasibility, accuracy (e.g., correlation, sensitivity, specificity) and acceptability of self-performed versus clinician-performed tests for vaginitis in adolescent females.

Approximately 300 adolescent females will undergo self- and clinician-testing for both STI and non-STI vaginitis. Subjects will be randomized into two groups. Group 1 will perform self-testing for the first half of the study before receiving clinician-testing for the remainder of the study. Group 2 participants will receive clinician-testing for the first half of the study before performing self-testing for the remainder of the study. All participants will have a discussion with the clinician to compare the results of self-performed tests with the results obtained by the clinician. Investigators will assess their acceptance of self- and clinician-testing before testing, after testing, and after the discussion with the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Sexual intercourse in the last 6 months
* Agree to perform self-testing
* Agree to pelvic examination

Exclusion Criteria:

* Have taken antibiotics used to treat vaginal infections in the 2 weeks prior to study entry or have used vaginal creams or medications in the 2 weeks prior to study entry

Ages: 14 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of self performed rapid trichomonas tests | Throughout study

SECONDARY OUTCOMES:
Acceptability of self testing for trichomonas | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Huppert, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Huppert JS, Mortensen JE, Reed JL, Kahn JA, Rich KD, Miller WC, Hobbs MM. Rapid antigen testing compares favorably with transcription-mediated amplification assay for the detection of Trichomonas vaginalis in young women. Clin Infect Dis. 2007 Jul 15;45(2):194-8. doi: 10.1086/518851. Epub 2007 Jun 6. PMID 17578778